CLINICAL TRIAL: NCT00142545
Title: Long-Term Safety and Effectiveness of Subcutaneous Injections of Apomorphine in the Treatment of "Off" Episodes in Patients With "On-Off" or "Wearing-Off" Effects Associated With Late-Stage Parkinson's Disease
Brief Title: Long Term Safety and Efficacy of SC Apomorphine in Treatment of "Off" Episodes in Late-Stage Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APO401
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2005-09-02 (Estimated); Status verified 2005-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

INTERVENTIONS:
Drug: apomorphine HCl injection

SUMMARY:
The current protocol is designed to satisfy the need for a compassionate use treatment protocol as well as for a long-term open label follow-up study.

DETAILED DESCRIPTION:
The primary objective of APO401 was to gain additional safety data in the outpatient use of apomorphine. APO401 provided an opportunity for all patients who had participated in a Mylan-sponsored placebo controlled trial of apomorphine to receive apomorphine therapy as ambulatory outpatients. Patients other than those enrolled in a Mylan-sponsored study were allowed to participate. Additional data regarding the safety and effectiveness of outpatient use of subcutaneous apomorphine were derived from this experience.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in a MYLAN sponsored study of subcutaneous apomorphine administration for the treatment of Off episodes due to end-of-dose motor deterioration ("Wearing-Off" effect) or sudden loss of mobility at seemingly random intervals ("On-Off" effect). With prior approval from MYLAN, patients other than those enrolled in a MYLAN sponsored study were allowed to participate. Following approval of Amendment 01, patients who met all other criteria for inclusion, regardless of previous participation in an apomorphine study, were allowed to participate.
* Age: Adults of any age > 18.
* Sex: Men and non-pregnant, non-lactating women.
* Women of childbearing potential must have had a negative serum (Beta HCG) pregnancy test within 14 days of the study start.
* Women of childbearing potential must have used an acceptable form of contraception.
* Patients with a clinical diagnosis of idiopathic Parkinson's Disease, i.e., not induced by drugs or caused by other diseases.
* Patients classified as stage II - V of the Hoehn and Yahr scale for staging the severity of Parkinson's Disease.
* Patients with refractory motor fluctuations of any frequency or duration. These include but are not necessarily limited to patients with the following symptoms:

  * Immobility resulting from regular dose failures.
  * Severe Off period discomfort.
  * Nocturnal/early morning dystonias.
  * Voiding dysfunctions.
  * Swallowing difficulties associated with Off periods.
  * Off period visual hallucinations.
  * Severe biphasic dyskinesia.
* The patient (or a caregiver) had to be able to recognize an Off state, and be sufficiently motivated to learn how to use the apomorphine injection to control these periods.
* The patient (or a caregiver) had to be able to maintain On-Off diaries.
* Unless otherwise specified, enrolled patients must be on an optimally maximized oral therapy regimen. Optimized oral anti-PD medication included: levodopa/carbidopa in either immediate or delayed release forms, plus at least one direct acting oral dopamine agonist for at least 30 days prior to enrollment into study.

Exclusion Criteria:

* Patients under medical therapy for clinically significant psychoses or dementia not related to ingestion of anti-PD medications. (Patients with hallucinations or other central adverse reactions associated solely with anti-PD medications were not excluded.)
* Patients with a history of drug or alcohol dependency within one year prior to study enrollment.
* Patients with unstable and clinically significant disease of cardiovascular (including orthostatic hypotension), hematologic (including Coombs' positive hemolytic anemia), hepatic, renal, metabolic, respiratory, gastrointestinal or endocrinological systems or neoplasm within the three months before the start of the study.
* Patients with a history of true allergy to morphine or its derivatives (including apomorphine), sulfur, sulfur containing medication, sulfites, sulfates, Tigan(R) (trimethobenzamide).
* Patients treated with experimental agents (other than apomorphine intermittent subcutaneous injections) within 30 days before study entry. Patients with participation in Bertek-sponsored study APO202 were excluded from participation in this study.
* Patients whose apomorphine regimen was characterized by administration methods other than intermittent subcutaneous injection.
* Patients who could not or would not sign an Informed Consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 1999-07; Study Completion 2005-07

PRIMARY OUTCOMES:
adverse events (AE)s
clinical laboratory tests
vital signs
electrocardiogram
orthostatic monitoring

SECONDARY OUTCOMES:
• Hoehn and Yahr Score
• UPDRS score - Motor Exam (Section III)
• UPDRS score - Total
• UPDRS score - Non-Motor Exam (Subtotal of Sections I, II, and IV)
• UPDRS score - Complications of Therapy (Section IV)
• Number of Off episodes based diary entries
• Duration of Off episodes based on diary entries
• Number of daily injections based on diary entries
• Length of time from injection to On based on diary entries

CONTACTS AND LOCATIONS:
Overall Officials: Will Sullivan, Study Director — Mylan Bertek Pharmaceuticals
Locations (1):
- Mylan Pharmaceuticals, Morgantown, West Virginia, United States